CLINICAL TRIAL: NCT07173140
Title: A Two Site Pilot Study of Functional and Microstructural Imaging Using Magnetic Resonance Imaging in Patients With Renal Tumours
Brief Title: Renal Tumour Imaging Using MRI
Acronym: RIM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other); University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 162190
Record Dates: First submitted 2025-08-18; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Renal Cancer; MRI; Small Renal Mass; Kidney Cancers
Keywords: Renal cancer; MRI; Small Renal Mass; Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Masking Description: Scan readers are blinded to lesion histology at the time of region of interest (ROI) drawing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Histological characterisation of renal tumours (No Intervention): Histological samples of ten patients with tumour histology will be retreived from the Royal Free Hospital Biobank. Slides will be stained using H&E and CD34 and cell size, stromal space and vascularity will be estimated and used to inform diffusion weighted imaging models.
- Comparison of microstructural MRI to histology (Experimental): 10 patients with small renal tumours will undergo microstructural MRI. Following MRI the tumours will be surgically resected. The MRI will be co-registered with histology. The degree of correlation between the MRI and underlying histology will be determined.
  Interventions: Diagnostic Test: MRI
- Repeatability of MRI of small renal masses (Experimental): The repeatability of the MRI scan of the small renal mass will be determined by participants undergoing a repeat MRI examination shortly after the first (within 14 d) on the same scanner.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Participants undergo an additional MRI scan using novel MRI sequences
  Arms: Comparison of microstructural MRI to histology; Repeatability of MRI of small renal masses

SUMMARY:
This study investigates whether new types of MRI scans can tell the difference between different kidney tumours before surgery. Currently, imaging scans can detect kidney tumours and their size, but they aren't effective at determining the tumour type or its aggressiveness. Biopsies are an option, but they are invasive and may miss important cancerous cells. The aim is to use imaging to determine which tumours are aggressive so they can be treated early while avoiding unnecessary treatment of benign tumours.

Patients with small renal tumours (≤ 7 cm) who meet the other inclusion and exclusion criteria will be asked to have an additional MRI scan at University College London Hospital prior to surgery.

The imaging findings will be compared to the histology result from the removed tumour. In 10 patients the histology will be targeted to a specific location in the tumour based on the imaging. 10 patients will undergo a repeat MRI <14 d apart to test whether the MRI scans can give the same answer twice (the test repeatability).

The study is expected to run for 24 months and is funded by NIHR.

The chief investigator for the study is Dr Richard Hesketh (rhesketh@ucl.ac.uk).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and over
2. Confirmed renal tumour ≤ 7 cm planned for surgical resection
3. Willing and able to provide written informed consent
4. Able to lie supine for the duration of an MRI

Exclusion Criteria:

1. Contraindication to MRI e.g., cardiac pacemaker
2. Contraindication to MR contrast agents
3. Pregnancy
4. Breastfeeding
5. Deranged renal function (eGFR <30) in the last three months.
6. Previous treatment of the renal tumour e.g., ablation, radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of proton density fat fraction (PDFF) to differentiate different histological subtypes of renal tumours. | 1 year
  PDFF mean values will be calculated for each tumour in arms 2 and 3. Following surgery the means for each histological subtype will be calculated and tested for statistical significance.
Repeatability of proton density fat fraction (PDFF) measurements. | 1 year
  Participants in arm 3 will undergo repeat scanning with a short time interval between scans. The repeatability of PDFF measurements will be assessed using within subject standard deviation, repeatability coefficients and Bland-Altman analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Immediately

REFERENCES:
- [Derived] Sen S, Smith L, Caselton L, Clemente J, Tran M, Punwani S, Atkinson D, Hesketh RL, Panagiotaki E. Dual deep learning approach for non-invasive renal tumour subtyping with VERDICT-MRI. Npj Imaging. 2026 Jan 6;4(1):2. doi: 10.1038/s44303-025-00135-6. PMID 41495369

DOCUMENTS (1):
  • Study Protocol (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT07173140/Prot_000.pdf